CLINICAL TRIAL: NCT06261424
Title: IMPACT, a Supervised Rehabilitation Program for Spastic Ataxias: A Rater-blinded, Randomized Controlled Trial
Brief Title: Effects of a Supervised Rehabilitation Program on Disease Severity in Spastic Ataxias
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Chicoutimi (Other)
Collaborators: McGill University (Other); Université de Sherbrooke (Other); Université du Québec a Montréal (Other); Laval University (Other); University of Calgary (Other); Corporation de recherche et d'action sur les maladies héréditaires (CORAMH) (Unknown); Cégep de Jonquière (Unknown); Centre intégré universitaire de santé et de services sociaux du Saguenay-Lac-St-Jean (Unknown); Muscular Dystrophy Canada (Other); University of Alberta (Other); Integrated University Health and Social Services Center of the Capitale-Nationale (Other)
Responsible Party: Principal Investigator, Elise Duchesne, Full Professor, Université du Québec à Chicoutimi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-1426
Record Dates: First submitted 2023-12-21; First posted 2024-02-15 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Autosomal Recessive Spastic Ataxia of Charlevoix-Saguenay; Spastic Paraplegia 7
MeSH Terms: conditions — Spastic ataxia Charlevoix-Saguenay type; Spastic Paraplegia Type 7

STUDY DESIGN:
Intervention Model Description: A multicentre and controlled trial design.
Who Masked: Care Provider
Masking Description: All participants will be assessed at their respective neuromuscular clinic (Saguenay, Quebec, Montreal or Calgary) by physiotherapists trained according to standard operating procedures (SOP). These physiotherapists will not be involved in the supervision of the program and will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group will receive their usual care and will be asked to continue their usual activities and exercises for the whole project duration. Only one clinical guide exists for ataxia interventions and no specific guidelines for physiotherapy and occupational therapy interventions are specified in this guide in terms of frequency, duration and type of interventions that are effective with this population. Patients generally have an annual follow-up with a doctor or a clinical nurse at a Neuromuscular Diseases Clinic. Patients are then referred if needed for follow-up with the physiotherapist and occupational therapist. Typically, patients are referred to physiotherapy for mobility-related needs such as the introduction of a walking aid, orthotic and sometimes teaching an exercise program. In occupational therapy, patients are referred for needs such as the introduction of technical aids, home adaptation or the introduction of a wheelchair.
- Intervention group (Experimental): The intervention group will follow a 12-week rehabilitation program, 3 times a week (two sessions in a therapy room and one session of aquatherapy).
  Interventions: Procedure: IMPACT - rehabIlitation prograM for sPAstiC aTaxias

INTERVENTIONS:
Procedure: IMPACT - rehabIlitation prograM for sPAstiC aTaxias — The rehabilitation program will last 12 weeks and consists of three training sessions of 60 minutes per week (2 sessions in a therapy room and 1 session in an adapted pool with multiple levels of water) for a total of 36 sessions. Participants will be divided into 7 subgroups of 6 participants and each sub-group will be supervised by one physiotherapist (PT) and one physiotherapy technologist for safety considerations. It will focus on these three domains: 1) postural control; balance, trunk-limbs and multi-joints control and coordination and 3) functional mobility. Each domain contains a standardized list of exercises with different difficulty levels and specific times allocation. All exercises will be executed by the participants at each session at the appropriate difficulty level. The initial level of difficulty for each exercise will be determined by the PT based on individual results of the pre-intervention assessment and on individual performance, fatigue level and safety.
  Arms: Intervention group

SUMMARY:
Spastic ataxias are a group of diseases causing symptoms such as walking difficulties and balance impairments that lead to a high risk of falls. No pharmacological treatments exist to treat these diseases. Unfortunately, little effort is made to develop non-pharmacological treatments specific to spastic ataxias despite the detrimental impact of the disease on several aspects of an individual's life and the high cost of falls for society each year. The three objectives of this project are: 1) to determine the effect of a 12-week rehabilitation program on disease severity as compared with usual care for individuals with spastic ataxias; 2) to identify which factors can help (or not) the implementation of the program in the clinical settings ("reel world"); and 3) to explore the cost-benefits of IMPACT [rehabIlitation prograM for sPAstiC aTaxias]. The team has developed the program to specifically target symptoms present in these patients and was previously pilot-tested. Based on the results obtained in this pilot project, positive effects are expected concerning the disease severity of participants. The investigators want, with this project, provide to health care professionals an option to offer better-suited services to people living with spastic ataxia worldwide.

ELIGIBILITY:
Inclusion Criteria:

* have a confirmed genetic diagnosis of ARSACS or SPG7
* be able to maintain standing position and to transfert
* be authorized by their treating neurologist
* speak French or English
* be able to give informed consent.

Exclusion Criteria:

* have active participation in a rehabilitation program (self-reported information)
* have another condition causing physical limitations
* be uncomfortable in a swimming pool
* be pregnant.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Severity of ataxia | 64 weeks
  The severity of ataxia assessed using the Scale for the assessment and rating of Ataxia (SARA) has been chosen as the main variable based on several considerations. 1) it is one of the most widely used scales among recessive cerebellar ataxias in intervention studies, 2) it includes lower limbs motor impairments-induced mobility limitations items, 3) is significantly correlated with key impairments variables such as standing balance and walking speed, 4) and is a candidate for outcome measurement in foreseeable clinical trials.
  It has eight categories with accumulative score ranging from 0 (no ataxia) to 40 (most severe ataxia) It showed evidence of adequate content validity and excellent construct validity and internal consistency in ARSACS and we recently validated the French version.

SECONDARY OUTCOMES:
Medication change | 64 weeks
  Patients will be asked about the possibility of changing their medication. A list of medications will also be provided by the pharmacy.
Weight | 64 weeks
  Patients weight in kilograms
height | 64 weeks
  Patients height in meters
Physical activities | 64 weeks
  The Rapid Assessment of Physical Activity (RAPA) is a questionnaire used to assess physical activity levels.
  Each question has a 'Yes' or 'No' option. The total score of the first seven items is out of 7; participants choose which question corresponds to their activity level. Any score less than 6 is considered suboptimal. Strength training and flexibility are scored separately (strength training = 1, flexibility = 2, both = 3)
Walking speed. | 64 weeks
  The 10-meter walk test will be used to assess the short-distance walking speed at comfortable and maximum speeds. The validity and reliability of the 10mWT are both excellent in ARSACS (ICC = 0.99).
Standing balance | 64 weeks
  Berg balance scale will be used to assess balance and risk of falling. Its validity has been demonstrated in ARSACS.18 Participants' level of confidence in their balance will be assessed using the simplified balance confidence scale specific to daily activities
  It has 14 (0-4) categories with accumulative score ranging from 0 to 56. Interpretation: 0-20, wheelchair bound; 21-40, walking with assistance; 41-56, independent.
Balance confidence | 64 weeks
  Activities specific balance confidence-simplified (ABC-S) scale will aslo be use to assess balance (0-3 likert scale) This questionnaire includes 15 evaluation items, rated from 0 (not at all confident) to 3 (very confident), according to the person's confidence in maintaining their balance when performing various activities. The total score ranges from 0 (minimum confidence) to 45 (maximum confidence), and is obtained by adding together the scores for each item and converting them into a percentage.
Sitting balance | 64 weeks
  Sitting balance and trunk control will be assessed with the Ottawa sitting scale (OSS).
  The first six items are tested with the participant's feet on the ground ( /24) and the next six with the feet off the ground ( /24). The total score is calculated by adding together the scores for the two subsections (maximum score out of /48).
Activities of Daily Living | 64 weeks
  The Barthel Index will assess the level of independence in performing daily living activities.
Muscle tone | 64 weeks
  Lower limb muscle tone (spasticity) will be measured with the modified Ashworth scale.
  Score each muscle group evaluated according to the table below. *Scoring is performed within the available range of motion. 0: No increase in muscle tone. 1: Discrete increase in muscle tone manifested by a twitch followed by release or by minimal resistance at the end of the movement. 1+: Discrete increase in muscle tone manifested by a twitch followed by minimal resistance perceived over less than half the joint amplitude. 2: More marked increase in muscle tone affecting most of the joint amplitude, the joint being easily mobilized. 3: Significant increase in muscle tone making passive mobilization difficult. 4: Affected joint is fixed (no passive movement possible).
Life habits | 64 weeks
  The Assessment of Life Habits Questionnaire 4.0. (LIFE-H) was used to assess participation. It includes a total of 96 activities with one total score, two subscores (daily activities and social activities) and 12 domains divided equally between both subscores. For each activity, the level of accomplishment, type of assistance required and level of satisfaction are rated. Accomplishment includes the difficulty level and assistance required: a mean score of "0" refers to a complete disruption of participation (i.e. activity not accomplished), and "10" refers to full participation (i.e. activity accomplished without difficulty and assistance). The satisfaction level is measured on a 4-point scale, where a higher score indicates higher satisfaction ("4"). For the 3.0 version, a change of 0.5 (/9) is considered a minimal clinically important difference but is not documented for the version 4.0.
Community mobility | 7 consecutives days, 2 times
  The daily rest-activity pattern will be assessed using an ActiGraph wGT3X-BT activity monitor worn on the nondominant arm for 7 consecutive days before and after the intervention period. Intradaily variability and interdaily stability (IS), M10 (most active 10-hours), L5 (least active 5-hours), and relative amplitude (RA) will be derived using nonparametric rhythm analysis. The patient's perception of mobility limitations will be measured by the Life Space Assessment questionnaire.
Plasma | 64 weeks
  3 x 10ml EDTA tubes will be collected to obtain 6 x 0.5ml cryovials of plasma (protein)
DNA | 64 weeks
  3 x 10ml EDTA tubes will be collected to obtain 3 x 2ml cryovials of Buffy Coat (DNA).
Serum | 64 weeks
  3 x 5ml SST serum tubes will be collected to obtain 12 x 0.5ml serum (protein) cryovials.
RNA | 64 weeks
  3 PAXgene 2.5ml tubes (RNA) will be collected and frozen as is.
Urine | 64 weeks
  10 ml of urine will be collected and separated into 12 cryovials of 0.5 ml.
Saliva | 64 weeks
  12 ml of saliva will be collected to obtain 12 cryovials of 0.5 ml.
Mobility Life-space | 64 weeks
  Life-Space Assessment (LSA-F) is a 20-items questionnaire measures the extent of mobility, taking into account the person's interactions with the environment. It assesses mobility habits in five living environments: the rooms of the home (or living unit for people living in sheltered housing), the surroundings of the home (or living unit/housing environment), the neighborhood, the city and outside the city.
  Mobility area - Composite score, which is obtained by combining the level of mobility area achieved, the frequency of travel in each mobility area and the assistance required (technical aid and/or assistance of a person) to get there. The score ranges from 0 to 120, where 120 corresponds to an unrestricted mobility area.
Ataxia impact scale | 64 weeks
  Person-reported ataxia impact scale (PRAIS) is self-administered questionnaire consists of 38 questions and aims to understand the impact of ataxia on daily life. A score out of 100 results.
Lower limb coordination | 64 weeks
  It will be measured using the Lower Extremity Motor Coordination Test. It is a reliable tool in ARSACS (ICC = 0.82-0.99).
Peak respiratory flow and cough | 64 weeks
  Peak expiratory flow (PEF) is the maximum speed at which air can be expelled from the lungs during forced expiration.
Fatigue | 64 weeks
  Fatigue will be assess with the Fatigue Severity Scale (FSS) This scale is a method of assessing the impact of fatigue on the subject. It is a short questionnaire that assesses the level of fatigue. The questionnaire contains nine statements that assess the severity of fatigue symptoms on a 7-level likert scale and produce a score between 9 and 63. A high score is a sign of fatigue
Falls. | 64 weeks
  The fall history with and without injury will be self-reported according to the recommendations of the group of Elley et al. Participants will have to complete every day a fall logbook and a research assistant will contact them each month to document the circumstances and consequences of falls including injuries and medical consultations.
Patient-reported impression of change. | 64 weeks
  The patients-global impression of change will be used (3 questions, 7-level Likert self-reported scale) to assess the impression of change.It is sensitive to change. This questionnaire gives the patient's perception. The higher the score, the worse the situation.
Anxiety and Depression | 64 weeks
  Hospital Anxiety and Depression scale will assess anxiety and Depression
  The HADS is a screening instrument for anxiety and depressive disorders. It comprises 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven to depression (total D), giving two scores (maximum score for each = 21).
Pain characteristics | 64 weeks
  Brief Pain Inventory Short Form
Functional lower extremity strength | 64 weeks
  The 30CST is a measurement that assesses functional lower extremity strength. The total number of correctly performed sit-to-stand repetitions is counted. If the participant is more than halfway upright when the 30 seconds have elapsed, count this as a repetition. If the participant is unable or unwilling to perform the test correctly, enter "0 repetitions" for each trial on the scoring sheet. The validity of the result of each test must be entered on the scoring sheet (valid or invalid).
Focus group with intervention group participants | 1 day
  Each participant will take part in one focus group after the rehabilitation program. Also, a semi-structured interview guide covering the 7 dimensions of the TFA will be used.
Focus groups with stakeholders | 12 weeks
  One focus group per site will be conducted before and after the intervention. In addition, during the rehabilitation program, each PT will be asked to fill out a journal of observations every week that includes the CFIR intervention items. In addition, the Determinant of Implementation Behavior. Questionnaire will be administered to PT and assistants at T0 and T3.
Lower limb muscle activation | 64 weeks
  It will be measured using surface EMG. Surface myoelectric signals will be recorded at 2000 HZ using a 16-channel wireless system (Trigno™ EMG, Delsys, MA, USA).
Quality of life | 64 weeks
  Quality of life will be assessed with SF-12 is a generic questionnaire that assesses health-related quality of life from the participant's point of view. It can be self-administered or completed during an interview. It comprises 12 assessment items, divided into 7 domains. The scoring system provides two quality-of-life scores (0 to 100: poor to excellent), i.e., a subtotal for mental and social quality of life (MCS) and a subtotal for physical quality of life (PCS).
CBA analyses and Willingness to pay | 64 weeks
  Estimating the costs related to the use of health services, falls with and without injuries, and improvement in quality of life and our health indicators (main and secondary outcomes). Using data collected in medical records and the hospitalization data, we will use different variables to take into account the use of health services such as: 1) visits physicians or health care professionals; 2) home visits by home-care professionals; and 3) emergency or hospital stays. We will also use the project's information relative to the cost of the rehabilitation program such as: 1) the number of hours of assessments and supervision of the program/type of professional and 2) the hourly rate of professionals. The cost of setting up a rehabilitation program will be estimated by combining human and material resources.
Gait's temporal parameters | 64 weeks
  The GAITRite system is a 14ft carpet containing sensors activated by pressure exerted by the feet and providing x and y coordinates. Then, the footprint analysis can provides the gait temporal parameters such as step time, step length, cadence and speed.
Stance balance | 64 weeks
  Force platform
Postural balance | 64 weeks
  Postural balance will be assess with the wobble chair. This test measures the postural balance of the trunk during a balance task in a seated position on an unstable chair, where only movements of the lumbar spine are allowed to restore balance.

CONTACTS AND LOCATIONS:
Overall Officials: Elise Duchesne, Ph D., Study Director — Université du Québec à Chicoutimi
Locations (5):
- Canada (5):
  - CIUSSS de la Capitale-Nationale, Hôpital de Baie-Saint-Paul, Baie-Saint-Paul, Quebec
  - CIUSSS de la Capitale-Nationale, Hôpital de La Malbaie, La Malbaie, Quebec
  - CIUSSS du Centre-Sud-de-l'Île-de-Montréal, installation Centre de réadaptation Lucie-Bruneau, Montreal, Quebec
  - CIUSSS de la Capitale-Nationale, installation IRDPQ, Québec, Quebec
  - Clinique des maladies neuromusculaires du Centre intégré universitaire de santé et de services sociaux (CIUSSS) du Saguenay-Lac-Saint-Jean, installation Hôpital Jonquière, Saguenay, Quebec

IPD SHARING:
Plan to Share IPD: Yes
All information collected as part of this research project, as research data including biological material, will be stored securely in the data bank Banque de données et de matériel biologique des maladies neuromusculaires et autres maladies et conditions apparentées (BDMB-MNM-MCA).
  All research data of participants, including biological material, will be used by researchers to carry out research projects on neuromuscular and related diseases.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The research data will be kept for as long as it is useful for the advancement of scientific knowledge. These data will be share of other researchers around the world.
Access Criteria: All these research projects will first be evaluated and approved by the Research Ethics Committee : Comité de recherche du Centre intégré universitaire de santé et de services sociaux du Saguenay-Lac-Saint-Jean. Also, this commitee make the follow-up for these research projects.
  The principal investigator of this research will respect privacy and confidentiality regulations in Quebec and in Canada for any sharing data research with other authorized persons in any countries.

REFERENCES:
- [Background] Lessard I, Masterman V, Cote I, Gagnon C, Duchesne E. A rehabilitation program to increase balance and mobility in ataxia of Charlevoix-Saguenay: An exploratory study. PLoS One. 2022 Dec 28;17(12):e0279406. doi: 10.1371/journal.pone.0279406. eCollection 2022. PMID 36576926